CLINICAL TRIAL: NCT01274663
Title: A Phase 1 Placebo-Controlled Study To Assess The Safety, Tolerability, And Pharmacokinetics Of PF-05175157 After Administration Of Single Escalating Oral Doses Under Fasted And Fed Conditions In Healthy Volunteers
Brief Title: A Study Of PF-05175157 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B1731001
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Single Ascending Dose; Phase 1; Safety and Tolerability; PK; Healthy Subjects
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 10 mg PF-05175157 or Placebo (Experimental): Subjects will receive one dose of PF-05175157 or one dose of Placebo (2:1 ratio) in random order.
  Interventions: Drug: PF-05175157 or Placebo
- 30 mg PF-05175157 or Placebo (Experimental): Subjects will receive one dose of PF-05175157 or one dose of Placebo (2:1 ratio) in random order.
  Interventions: Drug: PF-05175157 or Placebo
- 100 mg PF-05175157 or Placebo (Experimental): Subjects will receive one dose of PF-05175157 or one dose of Placebo (2:1 ratio) in random order.
  Interventions: Drug: PF-05175157 or Placebo
- 300 mg PF-05175157 or Placebo (Experimental): Subjects will receive one dose of PF-05175157 or one dose of Placebo (2:1 ratio) in random order.
  Interventions: Drug: PF-05175157 or Placebo
- 600 mg PF-05175157 or Placebo (Experimental): Subjects will receive one dose of PF-05175157 or one dose of Placebo (2:1 ratio) in random order.
  Interventions: Drug: PF-05175157 or Placebo
- 800 mg PF-05175157 or Placebo (Experimental): Subjects will receive one dose of PF-05175157 or one dose of Placebo (2:1 ratio) in random order.
  Interventions: Drug: PF-05175157 or Placebo
- xxx mg PF-05175157 or Placebo (Experimental): Subjects will receive one dose of PF-05175157 or one dose of Placebo (2:1 ratio) in random order.
  Interventions: Drug: PF-05175157 or Placebo

INTERVENTIONS:
Drug: PF-05175157 or Placebo — One dose of PF-05175157 will be administered as a powder-in-capsule in the fasting state in the AM; correspondingly, one dose of a matched powder-in-capsule placebo will be administered in the fasting state in the AM.
  Arms: 10 mg PF-05175157 or Placebo
Drug: PF-05175157 or Placebo — One dose of PF-05175157 will be administered as a powder-in-capsule in the fasting state in the AM; correspondingly, one dose of a matched powder-in-capsule placebo will be administered in the fasting state in the AM.
  Arms: 30 mg PF-05175157 or Placebo
Drug: PF-05175157 or Placebo — One dose of PF-05175157 will be administered as a powder-in-capsule in the fasting state in the AM; correspondingly, one dose of a matched powder-in-capsule placebo will be administered in the fasting state in the AM.
  Arms: 100 mg PF-05175157 or Placebo
Drug: PF-05175157 or Placebo — One dose of PF-05175157 will be administered as a powder-in-capsule in the fasting state in the AM; correspondingly, one dose of a matched powder-in-capsule placebo will be administered in the fasting state in the AM.
  Arms: 300 mg PF-05175157 or Placebo
Drug: PF-05175157 or Placebo — One dose of PF-05175157 will be administered as a powder-in-capsule in the fasting state in the AM; correspondingly, one dose of a matched powder-in-capsule placebo will be administered in the fasting state in the AM.
  Arms: 600 mg PF-05175157 or Placebo
Drug: PF-05175157 or Placebo — One dose of PF-05175157 will be administered as a powder-in-capsule in the fasting state in the AM; correspondingly, one dose of a matched powder-in-capsule placebo will be administered in the fasting state in the AM.
  Arms: 800 mg PF-05175157 or Placebo
Drug: PF-05175157 or Placebo — One dose of PF-05175157 will be administered as a powder-in-capsule immediately after breakfast; correspondingly, one dose of a matched powder-in-capsule placebo will be administered immediately after breakfast.
  Arms: xxx mg PF-05175157 or Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of single oral doses of PF-05175157 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non child-bearing potential) subjects between the ages of 18 and 45 years (inclusive).
* Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurements, 12-lead ECG and clinical laboratory tests.
* In addition, subjects must have normal chest x-ray, normal pulmonary function tests and normal ophthalmological examination.
* Body Mass Index (BMI) of 17.5 to 29.5 kg/m2; and a total body weight > 50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies).
* Evidence or history of any chronic ongoing or current pulmonary disease.
* History of smoking in the past 5 years or history or evidence of habitual use of other (non-smoked) tobacco or nicotine-containing products within 3 months of Screening or positive cotinine test at Screening or Day 0.
* Active ocular disease including infection, glaucoma, seasonal allergies, dry-eye symptoms or retinal/optic nerve disease.
* Evidence or history of 'dry eye-syndrome', Meibomian gland disease, ocular inflammation (eg, uveitis, iritis), chronic blepharitis, any eye surgery including Lasik, any mechanical injury or chemical exposure to the ocular surface, use of ocular lubricants, or use of contact lenses.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of escalating single doses of PF-05175157 in healthy subjects | 5 months
Single dose pharmacokinetics of PF-05175157 | 5 months

SECONDARY OUTCOMES:
Exploratory pharmacodynamic biomarkers | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, South Miami, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1731001&StudyName=A%20Study%20Of%20PF-05175157%20In%20Healthy%20Volunteers